CLINICAL TRIAL: NCT03615183
Title: A Single-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Anti-Retroviral Activity of MK-8527 Monotherapy in Anti-Retroviral Therapy (ART)-Naïve, HIV-1 Infected Participants
Brief Title: A Study of MK-8527 in Human Immunodeficiency Type 1 Virus (HIV-1) Infected Participants (MK-8527-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8527-002; 2018-001861-18 (EudraCT Number); MK-8527-002 (Other: Merck Study Number)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Human Immunodeficiency Virus; AIDS Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Panel A: 10 mg MK-8527 (Experimental): Single oral dose of 10 mg MK-8527 capsule after an 8-hour fast
  Interventions: Drug: MK-8527
- Panel B: 3 mg MK-8527 (Experimental): Single oral dose of 3 mg MK-8527 capsule after an 8-hour fast
  Interventions: Drug: MK-8527
- Panel C: 1 mg MK-8527 (Experimental): Single oral dose of 1 mg MK-8527 capsule after an 8-hour fast. Dose level determined by results of previous panels.
  Interventions: Drug: MK-8527
- Panel D: ≤50 mg MK-8527 (Experimental): Single oral dose of ≤50 mg MK-8527 capsule after an 8-hour fast. Dose level determined by results of previous panels.
  Interventions: Drug: MK-8527
- Panel E: ≤50 mg MK-8527 (Experimental): Single oral dose of ≤50 mg MK-8527 capsule after an 8-hour fast. Dose level determined by results of previous panels.
  Interventions: Drug: MK-8527

INTERVENTIONS:
Drug: MK-8527 — Single oral capsule

SUMMARY:
This study will evaluate the anti-retroviral activity of MK-8527 in HIV-1 infected, ART-naïve participants. The primary hypothesis is that MK-8527 has superior anti-retroviral activity compared to placebo, as measured by change from baseline in plasma HIV-1 ribonucleic acid (RNA) at 168 hours postdose.

DETAILED DESCRIPTION:
Up to five panels (Panels A-E) of 6 participants each will be enrolled in a sequential manner. In each panel, participants will receive a single dose of MK-8527 up to 50 mg. Historical data from previous single does studies will be used for placebo (control) comparisons.

ELIGIBILITY:
Inclusion Criteria

* Other than HIV infection, is in good health
* Is documented HIV-1 positive
* Diagnosed with HIV-1 infection ≥ 3 months prior to screening or perform the French 2008 Haute Autorité de Santé (HAS) Algorithm to confirm chronic HIV.
* Is ART-naïve which is defined as having never received any antiretroviral agent or the following: ≤30 consecutive days of an investigational antiretroviral agent, excluding an Nucleoside reverse transcriptase inhibitors (NRTI), or ≤60 consecutive days of combination ART not including an NRTI
* Has not received an investigational agent or marketed ART within 30 days of study drug administration
* Is willing to receive no other ART for the monitoring period of the study
* Has a Body Mass Index (BMI) ≤35 kg/m^2, inclusive
* If the male participant has a female partner(s) of childbearing potential, he must agree to use a medically acceptable method of contraception during the study and for 120 days after the last dose of study drug. If their partner is pregnant, males must agree to use a condom and no additional method of contraception is required for the pregnant partner
* If the participant is a female with reproductive potential, she must demonstrate a serum β-human chorionic gonadotropin (β-hCG) level consistent with the nongravid state at the prestudy (screening) visit and agree to use (and/or have their partner use) 2 acceptable methods of birth control beginning at the prestudy (screening) visit, throughout the study (including washout intervals between treatment periods/panels) and until 28 days after the last dose of study drug.
* If the participant is a postmenopausal female: she is without menses for at least 1 year and have a documented follicle stimulating hormone (FSH) level in the postmenopausal range at prestudy (screening)
* If the participant is a surgically sterile female: she is status posthysterectomy, or oophorectomy

Exclusion Criteria

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases. Participants with a remote history of uncomplicated medical events (eg, uncomplicated kidney stones, as defined as spontaneous passage and no recurrence in the last 5 years, or childhood asthma) may be enrolled in the study at the discretion of the investigator.
* Is mentally or legally incapacitated at the time of the prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder over the last 5 years. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator.
* History of cancer (malignancy)
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Positive for hepatitis B surface antigen
* History of chronic hepatitis C unless there has been documented cure and/or participant with a positive serologic test for hepatitis C virus (HCV) has a negative HCV viral load (VL)
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks
* Unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study, until the poststudy visit.
* Participated in another investigational study within 4 weeks
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day.
* Consumes excessive amounts, defined as greater than 6 servings (1 serving approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Is an excessive smoker (i.e., more than 10 cigarettes/day) and is unwilling to restrict smoking to ≤10 cigarettes per day
* Has a positive urine drug screen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Matei Bals Infectious Diseases Institute ( Site 0001), Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Anti-retroviral therapy (ART)-naïve, participants with human immunodeficiency type 1 virus (HIV-1) infection were enrolled in this study.
Groups:
- Panel A: MK-8527 10 mg: Single oral dose of 10 mg MK-8527 in capsule form after an 8-hour fast
- Panel B: MK-8527 3 mg: Single oral dose of 3 mg MK-8527 in capsule form after an 8-hour fast
- Panel C: MK-8527 1 mg: Single oral dose of 1 mg MK-8527 in capsule form after an 8-hour fast
Period: Overall Study
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg | Panel D: ≤50 mg MK-8527 | Panel E: ≤50 mg MK-8527
Started | 6 | 6 | 5 | 0 (Panel D was not conducted as the scientific study objectives were met in the conducted panels.) | 0 (Panel E was not conducted as the scientific study objectives were met in the conducted panels.)
Completed | 6 | 6 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Panels D and E were not conducted as the scientific study objectives were met in the conducted panels.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg | Panel D: ≤50 mg MK-8527 | Panel E: ≤50 mg MK-8527 | Total
Number analyzed (Participants) | 6 | 6 | 5 | 0 | 0 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.8 (2.3) | 33.3 (9.0) | 31.2 (5.6) |  |  | 31.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 |  |  | 3
  Male | 4 | 5 | 5 |  |  | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 |  |  | 0
  Not Hispanic or Latino | 6 | 6 | 5 |  |  | 17
  Unknown or Not Reported | 0 | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  |  | 0
  Asian | 0 | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 | 0 |  |  | 0
  White | 6 | 6 | 5 |  |  | 17
  More than one race | 0 | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma HIV-1 RNA
Description: Blood samples were taken to determine HIV-1 RNA levels at Predose (baseline) and 168 hours postdose. Data were fitted with a longitudinal data analysis (LDA) model containing fixed effects for treatment, time and treatment by time interaction, and a random effect for participant.The change from baseline in plasma HIV-1 RNA in participants administered MK-8527 was calculated and results were compared with historical placebo data.
Time Frame: Baseline and 168 hours postdose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Participants from Panels D and E were not analyzed because they were not enrolled in the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
log10 copies/mL | -1.39 [-1.78 to -0.99] | -1.66 [-2.06 to -1.27] | -0.95 [-1.38 to -0.52]
Statistical Analysis 1: Comparison: Panel A: MK-8527 10 mg; It was hypothesized that the true mean difference in the plasma HIV-1 RNA reduction from baseline between MK- 8527 and placebo is at least 1.0 log10 copies/mL; Test type: Superiority — Adjusted by Placebo data pooled from historical placebo data from recent monotherapy studies in HIV-1 infected participants (NCT00100048, NCT01466985, NCT01152255, and NCT01353898) and fitted with a longitudinal data analysis (LDA) model containing fixed effects for study and time, and a random effect for participants; Posterior Mean Difference = -1.36 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8527 and placebo ≤ -1.0 copies/mL was 99.72%
Statistical Analysis 2: Comparison: Panel B: MK-8527 3 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Adjusted by Placebo data pooled from historical placebo data from recent monotherapy studies in HIV-1 infected participants (NCT00100048, NCT01466985, NCT01152255, and NCT01353898) and fitted with a LDA model containing fixed effects for study and time, and a random effect for participants; Posterior Mean Difference = -1.63 — PP of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8527 and placebo ≤ -1.0 copies/mL was 99.86%
Statistical Analysis 3: Comparison: Panel C: MK-8527 1 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; Posterior Mean Difference = -0.92 — PP of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8527 and placebo ≤ -1.0 copies/mL was 9.42%

2. Primary Outcome: Percentage of Participants Who Report 1 or More Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it is considered related to the medicinal product. The percentage of participants that reported at least 1 AE will be summarized.
Time Frame: Up to 28 days
Population: Participants who received at least one dose of the investigational drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
Percentage of participants | 0 | 33.3 | 0

3. Primary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to an AE
Description: An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it is considered related to the medicinal product. The percentage of participants that were discontinued from the study due to an AE will be summarized.
Time Frame: Up to 28 days
Population: Participants who received at least one dose of the investigational drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
Percentage of participants | 0 | 0 | 0

4. Secondary Outcome: Area Under the Concentration Time Curve From Hour 0 to 168 Hours (AUC0-168) of MK-8527-TP in Peripheral Blood Mononuclear Cells (PBMC)
Description: Blood samples were taken at Predose, up to 168 hours postdose to determine the AUC0-168 of MK-8527-triphosphate (MK-8527-TP) in PBMCs. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% confidence intervals (CI) for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*pmol/10^6 cells
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
hr*pmol/10^6 cells | 178 [140 to 226] | 64.1 [50.5 to 81.3] | 29.1 [22.4 to 37.7]

5. Secondary Outcome: Area Under the Concentration Time Curve From Hour 0 to Last (AUC0-last) of MK-8527-TP in PBMC
Description: Blood samples were taken at Predose, up to approximately 28 days postdose to determine the AUC0-last of MK-8527-TP in PBMCs. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 240, 336, 504, 672 hours or 28 days postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*pmol/10^6 cells
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
hr*pmol/10^6 cells | 235 [182 to 302] | 108 [84 to 139] | 49.5 [37.5 to 65.3]

6. Secondary Outcome: Area Under the Concentration Time Curve From Hour 0 to Infinity (AUC0-inf) of MK-8527-TP in PBMC
Description: Blood samples were taken at Predose, up to approximately 28 days postdose to determine the AUC0-Inf of MK-8527-TP in PBMCs. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 240, 336, 504, 672 hours or 28 days postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*pmol/10^6 cells
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
hr*pmol/10^6 cells | 265 [206 to 342] | 146 [113 to 188] | 55.0 [41.6 to 72.8]

7. Secondary Outcome: Maximum Concentration (Cmax) of MK-8527-TP in PBMC
Description: Blood samples were taken at Predose, up to approximately 28 days postdose to determine the Cmax of MK-8527-TP in PBMCs. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 240, 336, 504, 672 hours or 28 days postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
pmol/10^6 cells | 1.81 [1.40 to 2.35] | 0.644 [0.497 to 0.834] | 0.265 [0.200 to 0.352]

8. Secondary Outcome: Time to Cmax (Tmax) of MK-8527-TP in PBMC
Description: Blood samples were taken at Predose, up to approximately 28 days postdose to determine the Tmax of MK-8527-TP in PBMCs. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 240, 336, 504, 672 hours or 28 days postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
Hours | 18.00 [12.00 to 24.00] | 24.00 [12.00 to 24.00] | 24.00 [12.00 to 96.63]

9. Secondary Outcome: Concentration at 168 Hours (C168) of MK-8527-TP in PBMC
Description: Blood samples were taken at 168 hours postdose to determine the C168 of MK-8527-TP in PBMCs. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: 168 hours postdose for each panel
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
pmol/10^6 cells | 0.509 [0.371 to 0.698] | 0.334 [0.244 to 0.458] | 0.0978 [0.0692 to 0.138]

10. Secondary Outcome: Apparent Terminal Half Life (t1/2) of MK-8527-TP in PBMC
Description: Blood samples were taken at Predose, up to approximately 28 days postdose to determine the t1/2 of MK-8527-TP in PBMCs. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 240, 336, 504, 672 hours or 28 days postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
Hours | 117.84 (35.00) | 188.66 (122.5) | 210.93 (14.62)

11. Secondary Outcome: Area Under the Concentration Time Curve From Hour 0 to 168 Hours (AUC0-168) of MK-8527 in Plasma
Description: Blood samples were taken at Predose, up to 168 hours postdose to determine the AUC0-168 of MK-8527 in plasma. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 168 hours postdose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. The 1 mg MK-8527 arm had insufficient data for one participant. Participants from Panels D and E were not analyzed because they were not enrolled in the study.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*μmol/L
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 4
hr*μmol/L | 0.926 [0.719 to 1.19] | 0.152 [0.118 to 0.196] | 0.0189 [0.0138 to 0.0258]

12. Secondary Outcome: Area Under the Concentration Time Curve From Hour 0 to Last (AUC0-last) of MK-8527 in Plasma
Description: Blood samples were taken at Predose, up to 168 hours postdose to determine the AUC0-last of MK-8527 in plasma. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*μmol/L
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
hr*μmol/L | 0.880 [0.669 to 1.16] | 0.121 [0.0919 to 0.159] | 0.0151 [0.0112 to 0.0204]

13. Secondary Outcome: Area Under the Concentration Time Curve From Hour 0 to Infinity (AUC0-inf) of MK-8527 in Plasma
Description: Blood samples were taken at Predose, up to 168 hours postdose to determine the AUC0-inf of MK-8527 in plasma. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 168 hours postdose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. The 1 mg MK-8527 arm had insufficient data for four participants. Participants from Panels D and E were not analyzed because they were not enrolled in the study.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*μmol/L
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 1
hr*μmol/L | 1.10 [0.794 to 1.53] | 0.196 [0.141 to 0.272] | NA [NA to NA] — NA was due to insufficient participants

14. Secondary Outcome: Maximum Concentration (Cmax) of MK-8527 in Plasma
Description: Blood samples were taken at Predose, up to 168 hours postdose to determine the Cmax of MK-8527 in plasma. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
μmol/L | 0.177 [0.114 to 0.276] | 0.0371 [0.0238 to 0.0577] | 0.0162 [0.00998 to 0.0264]

15. Secondary Outcome: Time to Cmax (Tmax) of MK-8527 in Plasma
Description: Blood samples were taken at Predose, up to 168 hours postdose to determine the Tmax of MK-8527 in plasma. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 168 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
Hours | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.50]

16. Secondary Outcome: Concentration at 168 Hours (C168) of MK-8527 in Plasma
Description: Blood samples were taken at 168 hours postdose to determine the C168 of MK-8527 in plasma. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 5
μmol/L | NA [NA to NA] — Results were below the lower limit of quantitation. | NA [NA to NA] — Results were below the lower limit of quantitation. | NA [NA to NA] — Results were below the lower limit of quantitation.

17. Secondary Outcome: Apparent Terminal Half Life (t1/2) of MK-8527 in Plasma
Description: Blood samples were taken at Predose, up to 168 hours postdose to determine the t1/2 of MK-8527 in plasma. Values were natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The 95% CI for the means were constructed on the natural log scale and referenced the t-distribution.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 168 hours postdose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
Number analyzed (Participants) | 6 | 6 | 1
Hours | 40.31 (60.27) | 12.36 (78.23) | NA (NA) — NA was due to insufficient participants

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Participants who received at least one dose of the investigational drug. Panels D and E were not conducted as the scientific study objectives were met in the conducted panels.
Arm/Group | Panel A: MK-8527 10 mg | Panel B: MK-8527 3 mg | Panel C: MK-8527 1 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-8527 10 mg (N=6) | Panel B: MK-8527 3 mg (N=6) | Panel C: MK-8527 1 mg (N=5)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT03615183/Prot_SAP_000.pdf